CLINICAL TRIAL: NCT06281691
Title: GreenBladder - Early Detection of Bladder Cancer in Residents in Greenland Using a Urinary Marker and a Mobile Cystoscopy Unit
Status: Enrolling by invitation | Type: Observational
Sponsor: Jørgen Bjerggaard Jensen (Other)
Collaborators: Cepheid (Industry); Laborie Medical Technologies Inc. (Industry); Vingmed Danmark A/S (Individual); OneMed A/S (Unknown)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: GreenBladder
Record Dates: First submitted 2024-01-30; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Greenlandic citizens aged 18 years and above, referred for cystoscopy: Patients who have been referred for a cystoscopy will be invited to participate in the study. During their cystoscopy appointment, they will be asked to provide a urine sample for the Xpert bladder cancer detection test.
  Interventions: Diagnostic Test: Xpert® Bladder Cancer Detection Test

INTERVENTIONS:
Diagnostic Test: Xpert® Bladder Cancer Detection Test — A urine sample is analyzed with the Xpert® Bladder Cancer Detection Test

SUMMARY:
The goal of this observational study is to evaluate whether a urinary biomarker (Xpert® Bladder Cancer Detection Test) can be used as a selection tool to decide which patients that should undergo cystoscopy in haematuria work-up or in other indications where bladder tumor is suspected. Hereby, the investigators will investigate in which patients where cystoscopy can be omitted, particularly in areas with limited access to urological service. With these more selected investigations, patients with bladder tumors will potentially be selected to earlier diagnosis compared to the current non-selected investigations with the inherent logistic and economical challenges. With this strategy, the investigators aim at improving the current poor prognosis for bladder cancer patients in Greenland.

DETAILED DESCRIPTION:
Methods:

Citizens of Greenland above the age of 18 years referred for cystoscopy will be invited to participate in an observational study at the time of already planned cystoscopy.

Hypothesis:

The investigators hypothesize that the Xpert® Bladder Cancer Detection test can identify patients with a bladder tumor and serve as a future selection tool to support clinical decision whether to perform a cystoscopy or not - especially in areas with limited access to urological services.

Perspectives:

The investigators hope to improve the current poor prognosis for bladder cancer patients in Greenland with the early detection. If this is successful, it could change the way patients are examined for bladder cancer in Greenland, but in the long term also in Denmark and other countries. Thus, the study will be able to determine whether a simple urine examination should be introduced early in the current cancer program in order to reduce the number of patients who need to undergo a cystoscopy and who can avoid this and get an earlier clarification.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of signing the Informed Consent Form with an indication for cystoscopy and planned for this already at study inclusion.
* Ability to understand the Participant Information Sheet orally and in writing in either Danish or Greenlandic.
* Signed Informed Consent Form.
* Is, according to the Investigator's judgement, able to comply with the trial protocol.

Exclusion Criteria:

* Patients not willing to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 and above who reside in Greenland and are currently on the waiting list to undergo cystoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of urinary marker (Xpert Bladder Cancer Detection Test) in patients undergoing cystoscopy for bladder cancer investigation | Baseline
  To assess the reliability and precision of Xpert Bladder Cancer Detection test ability to correctly identify cases of bladder cancer in patients as part of the diagnostic investigation

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie D Fryd, MD, Principal Investigator — PhD student
Locations (2):
- Department of Urology, Aarhus University Hopsital, Aarhus, Denmark
- Queen Ingrid's Hospital, Nuuk, Greenland

IPD SHARING:
Plan to Share IPD: No